CLINICAL TRIAL: NCT01607398
Title: A 12-week Randomised, Double-blind, Parallel-group Study to Evaluate the Anti-inflammatory Effects of ADOAIR® 50/250mcg Twice Daily Compared With Placebo Twice Daily in Japanese Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: ADOAIR250 Anti-inflammatory Effects in Japanese Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116571
Record Dates: First submitted 2012-05-10; First posted 2012-05-30 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Japan; COPD; CAT; placebo; serum; Adoair250; anti-inflammatory; sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADOAIR250 (Experimental): ADOAIR 250mcg inhalations, twice daily, from week0 - 12
  Interventions: Drug: ADOAIR250
- Placebo (Placebo Comparator): Placebo inhalation, twice daily, from week0 -12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADOAIR250 — 250 mcg inhalation, twice daily, from week0 -12.
  Arms: ADOAIR250
Drug: Placebo — Placebo inhalation, twice daily, from week0 -12.
  Arms: Placebo

SUMMARY:
The study will be conducted in a respiratory specialist institute in Japan, with standardized techniques and data assurance checks to optimize data quality. The licensed dosage and administration of Adoair in Japan will be applied in this study. Each subject will receive treatment options in a randomized blinded fashion. Subjects will be randomized following a 4-week wash-out phase to take either Adoair 50/250mcg twice daily or placebo twice daily for 12 weeks.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, two-arm, parallel-group, 12-week-treatment study in Japanese patients with COPD.

At Visit 1, patients confirmed to be fulfilling all the inclusion criteria and not meeting any of the exclusion criteria will start the 4-week run-in period. During the entire study period, including the run-in period, the only drug allowed to use in addition to the study drug will be oxitropium (short-acting anticholinergic drug) as relief medication. At the end of the run-in period (Visit 2), subjects eligible for randomisation will be evenly randomised to one of the following two treatment groups and start the 12-week treatment period.

* ADOAIR®250 one inhalation twice daily from the DISKUS inhaler
* Placebo one inhalation twice daily from the DISKUS inhaler

Study completers will be defined as subjects who have completed all examinations, assessments, and study procedures in the study period, including the run-in period and the follow-up period. At completion/discontinuation of the treatment period, subjects will be switched to appropriate COPD treatment at the discretion of the investigator (or subinvestigator).

ELIGIBILITY:
Inclusion Criteria:

1. Japanese (male or female) outpatients aged 40-80 years inclusive at Visit 1 (Female patients may be enrolled only if they are not of child-bearing potential, or are of child-bearing potential who agree to properly use protocol-specified contraceptive measures. )
2. Have a diagnosis of COPD (defined as per the COPD guideline)
3. Have a FEV1/FVC ratio < 0.70 at 15-60 minutes following use of SALTANOL® INHALER
4. Have a FEV1 of >= 40% to < 80% of the predicted normal value at 15-60 minutes following use of SALTANOL® INHALER
5. Current or ex-smokers with a smoking history of at least 10 pack-years
6. Able to use the DISKUS inhaler and the short-acting inhaled anticholinergic drug
7. Capable of providing written voluntary consent to participate in the study

Exclusion Criteria:

1. Diagnosed by the investigator (or subinvestigator) as having bronchial asthma
2. Have any respiratory disorder other than COPD (e.g., lung cancer, sarcoidosis, tuberculosis [including old tuberculosis], pulmonary fibrosis)
3. Have a chest X-ray (or CT scan) indicating a diagnosis other than COPD that might interfere with assessments in the study (This must be assessed using last imaging study performed within 6 months prior to Visit 1; or, a chest X-ray must be obtained at Visit 1.)
4. Have chronic respiratory failure
5. Have undergone lung volume reduction and/or lung transplant
6. Have had a COPD exacerbation or respiratory infection requiring systemic corticosteroid or microbial therapy or hospitalisation, within 6 weeks prior to Visit 1
7. Have used inhaled corticosteroids and systemic corticosteroids within 4 weeks prior to Visit 1
8. Have used long-acting β2 agonists (inhaled or patch) within 2 weeks prior to Visit 1
9. Are unable to stop their short-acting β2 agonist therapy at Visit 1 (During the study participation, oxitropium bromide (TERSIGAN) will be used as relief medication.)
10. Receiving long-term oxygen therapy with oxygen use for more than 12 hours per day
11. Have a concurrent serious or uncontrolled disease that might interfere with assessments in the study (including psychiatric disease, unstable liver disease, and heart disease)
12. Have a QTc > 450 msec (or > 480 msec in patients with bundle branch block) at Visit 1 (based on average QTc from three consecutive cardiac cycles on ECG)
13. Have participated in another study and received any other study drug within 4 weeks prior to Visit 1
14. Diagnosed by the investigator (or subinvestigator) as having drug or alcohol dependence
15. Have known or suspected hypersensitivity to bronchodilators, inhaled corticosteroid, or lactose
16. Have known α1 antitrypsin deficiency
17. Previously enrolled in this study
18. Judged by the investigator (or subinvestigator) to be inappropriate to participate in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Osaka, Japan

REFERENCES:
- [Derived] Asai K, Kobayashi A, Makihara Y, Johnson M. Anti-inflammatory effects of salmeterol/fluticasone propionate 50/250 mcg combination therapy in Japanese patients with chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2015 Apr 17;10:803-11. doi: 10.2147/COPD.S79842. eCollection 2015. PMID 25945045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese participants with Chronic Obstructive Pulmonary Disease (COPD) were enrolled in this study.
Pre-assignment Details: At Visit 1, participants meeting the inclusion criteria and not meeting any of the exclusion criteria entered a 4-week Run-in Period. At the end of the Run-in Period (Visit 2), eligible participants were randomized to a 12-week Treatment Period.
Groups:
- Placebo: Participants self-administered one inhalation of placebo powder twice daily from a dry powder inhaler for 12 weeks. Participants used oxitropium (a short-acting anticholinergic drug) as a relief medication during the study.
- ADOAIR 250: Participants self-administered one inhalation of ADOAIR 250 (salmeterol 50 micrograms [µg] and fluticasone propionate 250 µg) powder twice daily from a dry powder inhaler for 12 weeks. Participants used oxitropium (a short-acting anticholinergic drug) as a relief medication during the study.
Period: Overall Study
Arm/Group | Placebo | ADOAIR 250
Started | 28 | 28
Completed | 26 | 26
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Severe COPD | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ADOAIR 250 | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data are reported for members of the Per Protocol Population, comprised of all participants who had an evaluable sputum sample at Baseline and at the endpoint of interest, were randomized to study treatment and received at least one dose of study medication, and had no major protocol violations.
  Years | 62.2 (8.06) | 64.7 (9.31) | 63.4 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data are reported for members of the Per Protocol Population, comprised of all participants who had an evaluable sputum sample at Baseline and at the endpoint of interest, were randomized to study treatment and received at least one dose of study medication, and had no major protocol violations.
  Participants
    Female | 0 | 1 | 1
    Male | 26 | 25 | 51
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data are reported for members of the Per Protocol Population, comprised of all participants who had an evaluable sputum sample at Baseline and at the endpoint of interest, were randomized to study treatment and received at least one dose of study medication, and had no major protocol violations.
  participants
    Asian-Japanese Heritage | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Neutrophil Count in Induced Sputum at Week 12
Description: Induced sputum samples were collected at Baseline and at Week 12. The neutrophil count in induced sputum was measured with the use of a cytological specimen of inflammatory cells in the induced sputum. Change from Baseline in neutrophil count was calculated as the Week 12 value minus the Baseline value (percentage of neutrophil of total cells in induced sputum at Week 12 minus the Baseline value).
Time Frame: Baseline and Week 12
Population: Per Protocol Population: all participants who had an evaluable sputum sample at Baseline and at the endpoint of interest, were randomized to study treatment and received at least one dose of study medication, and had no major protocol violations. Only those participants available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: ratio (%)
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 21 | 24
ratio (%) | 1.35 [-15.50 to 6.30] | -6.00 [-30.50 to 6.90]
Statistical Analysis 1: Comparison: Placebo vs ADOAIR 250; Test type: Superiority or Other; p = 0.5146, Wilcoxon (Mann-Whitney); The analysis was done using the Van Elteren extension to the Wilcoxon rank sum test; Median Difference (Final Values) = -8.05, 95% CI 2-sided [-20.500 to 7.600] — From Van-Elteren extension to the Wilcoxon Rank Sum test, adjusted for smoking status strata and Hodges-Lehmann estimator of the 95% CI, not stratified and unadjusted for multiplicity

2. Secondary Outcome: Change From Baseline in All Inflammatory Cell Count in Induced Sputum at Week 12
Description: Induced sputum samples were collected at Baseline and at Week 12. All inflammatory cells in induced sputum were counted with the use of a cytological specimen of cells in the induced sputum. Change from Baseline in all inflammatory cell count was calculated as the Week 12 value minus the Baseline value.
Time Frame: Baseline and Week 12
Population: Per Protocol Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Cells per millimeters cubed (cells/mm^3)
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 25 | 24
Cells per millimeters cubed (cells/mm^3) | -0.0080 [-0.3560 to 0.1400] | -0.0280 [-0.3170 to 0.2255]

3. Secondary Outcome: Change From Baseline in Interferon (INF)-Gamma-positive Cells and Perforin-positive Cells in Sputum at Week 12
Description: INF-gamma-positive cells and perforin-positive cells were not detected in samples collected in this study due to the conditions of the samples and/or antibodies. No re-assays were performed, "no result"/"no data" was entered into the case report forms, and no statistical analysis or data summarization was performed.
Time Frame: Baseline and Week 12
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Interleukin (IL)-8 Levels in Sputum Supernatant at Week 12
Description: Induced sputum samples were collected at Baseline and at Week 12. The levels of IL-8 in the supernatant of an induced sputum sample were measured at the same time using the multiplex assay system. Change from Baseline in IL-8 levels was calculated as the Week 12 value minus the Baseline value.
Time Frame: Baseline and Week 12
Population: Per Protocol Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Picograms per milliliter (pg/mL)
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 25 | 25
Picograms per milliliter (pg/mL) | -5.0 [-177.00 to 267.20] | -30.0 [-1930.00 to 850.00]

5. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP) Levels in Sputum Supernatant at Week 12
Description: Data cannot be reported because hsCRP was under the lower limit of detection in all samples.
Time Frame: Baseline and Week 12
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Myeloperoxidase (MPO) and Pulmonary Surfactant Protein (SP)-D Levels in Sputum Supernatant at Week 12
Description: Induced sputum samples were collected at Baseline and at Week 12. The levels of MPO and SP-D in the supernatant of an induced sputum sample were measured at the same time using the multiplex assay system. Change from Baseline in MPO and SP-D levels was calculated as the Week 12 value minus the Baseline value.
Time Frame: Baseline and Week 12
Population: Per Protocol Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 25 | 25
ng/mL
  MPO | 1.80 [-227.30 to 49.80] | -23.90 [-157.20 to 33.10]
  SP-D | 0.00 [-17.30 to 7.80] | 0.00 [-19.10 to 42.00]

7. Secondary Outcome: Change From Baseline in IL-6 and IL-8 Levels in Serum at Week 12
Description: Serum samples were collected at Baseline and at Week 12. The levels of IL-6 and IL-8 in serum samples were measured at the same time using the multiplex assay system. Change from Baseline in IL-6 and IL-8 levels was calculated as the Week 12 value minus the Baseline value.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
pg/mL
  IL-6 | 0.30 [-0.10 to 1.40] | 0.35 [-0.40 to 1.00]
  IL-8 | -1.80 [-5.50 to 6.60] | -0.20 [-2.20 to 2.60]

8. Secondary Outcome: Change From Baseline in hsCRP, SP-D, and Clara Cell Protein 16 (CC 16) Levels in Serum at Week 12
Description: Serum samples were collected at Baseline and at Week 12. The levels of hsCRP, SP-D, and CC16 in serum samples were measured at the same time using the multiplex assay system. Change from Baseline in hsCRP, SP-D, and CC16 was calculated as the Week 12 value minus the Baseline value.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
ng/mL
  hsCRP | 107.0 [-143.0 to 653.0] | 23.5 [-90.0 to 460.0]
  SP-D | -0.10 [-15.70 to 11.0] | -0.20 [-7.90 to 4.60]
  CC-16 | -0.05 [-0.60 to 0.40] | -0.05 [-1.20 to 0.00]

9. Secondary Outcome: Change From Baseline in Fibrinogen Levels in Serum at Week 12
Description: Per Protocol Amendment 4, the measurement of fibrinogen levels in serum was removed from the analysis plan because fibrinogen levels were found to be too low and too difficult to measure.
Time Frame: Baseline and Week 12
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC) at Week 12
Description: FEV1 and FVC are measures of lung function. FEV1 is defined as the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. Respiratory function tests were performed for the measurement of FEV1 and FVC at Baseline and at Week 12. The values were measured at 15 to 60 minutes following the use of a pressurized metered-dose inhaler. Three technically acceptable values were obtained, and the highest value was recorded. Change from Baseline in FEV1 and FVC was calculated as the Week 12 value minus the Baseline value.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Median (Inter-Quartile Range); unit: Liters (L)
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Liters (L)
  FEV1 | 0.035 [-0.090 to 0.130] | 0.020 [-0.030 to 0.130]
  FVC | -0.035 [-0.130 to 0.170] | -0.055 [-0.250 to 0.190]

11. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Question 1 Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8) designed to assess the health status of participants with COPD. In Question 1, participants were asked to rate how much they cough on a scale of 0 to 5: 0, "I never cough"; 5, "I cough all the time." Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | 0.1 (0.89) | -0.5 (1.27)

12. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Question 2 Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8) designed to assess the health status of participants with COPD. In Question 2, participants were asked to rate the amount of phlegm (mucus) in their chest on a scale of 0 to 5: 0, "I have no phlegm (mucus) in my chest at all"; 5, "My chest is completely full of phlegm (mucus)." Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | -0.2 (1.33) | 0.0 (1.34)

13. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Question 3 Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8) designed to assess the health status of participants with COPD. In Question 3, participants were asked to rate how tight their chest feels on a scale of 0 to 5: 0, "My chest does not feel tight at all"; 5, "My chest feels very tight." Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | 0.2 (1.03) | 0.0 (1.41)

14. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Question 4 Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8) designed to assess the health status of participants with COPD. In Question 4, participants were asked to rate how breathless they feel when walking up a flight of stairs or a hill on a scale of 0 to 5: 0, "When I walk up a hill or one flight of stairs I am not breathless"; 5, "When I walk up a hill or one flight of stairs I am very breathless." Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | -0.7 (1.41) | 0.1 (1.11)

15. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Question 5 Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8) designed to assess the health status of participants with COPD. In Question 5, participants were asked to rate how limited they are in doing activities at home on a scale of 0 to 5: 0, "I am not limited doing any activities at home"; 5, "I am very limited doing activities at home." Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | 0.1 (1.11) | 0.0 (0.92)

16. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Question 6 Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8) designed to assess the health status of participants with COPD. In Question 6, participants were asked to rate how confident they are leaving home despite their lung condition on a scale of 0 to 5: 0, "I am confident leaving my home despite my lung condition"; 5, "I am not at all confident leaving my home because of my lung condition." Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | -0.1 (0.59) | 0.1 (0.93)

17. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Question 7 Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8) designed to assess the health status of participants with COPD. In Question 7, participants were asked to rate how soundly they sleep on a scale of 0 to 5: 0, "I sleep soundly"; 5, "I don't sleep soundly because of my lung condition." Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | 0.2 (1.08) | 0.0 (1.55)

18. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Question 8 Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8) designed to assess the health status of participants with COPD. In Question 8, participants were asked to rate how much energy they have on a scale of 0 to 5: 0, "I have lots of energy"; 5, "I have no energy at all." Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | -0.1 (0.89) | 0.2 (1.06)

19. Secondary Outcome: Change From Baseline in the COPD Assessment Test (CAT) Total Score at Week 12
Description: Participants completed the CAT questionnaire before undergoing respiratory function tests at Baseline and at Week 12. The CAT questionnaire is an 8-item questionnaire (comprised of Question [Q] 1 to Q8; each question scored from 0 to 5) designed to assess the health status of participants with COPD. The total score is calculated as the sum of the scores from Questions 1 to 8, for a range of possible scores of 0 to 40. A higher total score represents a lower quality of life, and vice versa. Change from Baseline was calculated as the Week 12 score minus the Baseline score.
Time Frame: Baseline and Week 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Scores on a scale | -0.5 (4.45) | -0.2 (4.18)

20. Secondary Outcome: Number of Participants Who Experienced the Indicated Number of COPD Exacerbations During the Treatment Period
Description: The occurrence of a COPD exacerbation was assessed on each day of evaluation during the treatment period per the defined severity classifications. COPD exacerbations were classified based on severity as a mild exacerbation (exacerbation of COPD symptoms were manageable by the participant, not requiring systemic corticosteroid or antimicrobial therapy), a moderate exacerbation (exacerbation of COPD symptoms required systemic corticosteroid or antimicrobial therapy), or a severe exacerbation (exacerbation of COPD symptoms required hospitalization). The number of participants who experienced 0, 1, 2, and >=3 exacerbation(s) was summarized.
Time Frame: From Baseline up to Week 12
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | Placebo | ADOAIR 250
Number analyzed (Participants) | 26 | 26
Participants
  0 moderate exacerbations | 25 | 26
  1 moderate exacerbation | 1 | 0
  2 moderate exacerbations | 0 | 0
  >=3 moderate exacerbations | 0 | 0
  0 severe exacerbations | 26 | 26
  1 severe exacerbation | 0 | 0
  2 severe exacerbations | 0 | 0
  >=3 severe exacerbations | 0 | 0
  0 overall exacerbations | 25 | 26
  1 overall exacerbation | 1 | 0
  2 overall exacerbations | 0 | 0
  >=3 overall exacerbations | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of administration of the study drug until the end of follow-up (approximately up to Week 13).
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | Placebo | ADOAIR 250
Serious Adverse Events (participants affected / at risk) | 2/28 | 1/28
Other Adverse Events (participants affected / at risk) | 12/28 | 14/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | ADOAIR 250 (N=28)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | ADOAIR 250 (N=28)
Nasopharyngitis (Infections and infestations) | 5 | 2
Oral candidiasis (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.